CLINICAL TRIAL: NCT00566072
Title: The Influence of Intensive Education and Coaching on Compliance for Oral Ganciclovir in the Prophylaxis of CMV: an Open Randomised Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Isabelle Devolder, University Hospital Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2001/181
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Cytomegalovirus Infections
Keywords: the effect of information on compliance of medication
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): instructions and coaching on the use and intake of ganciclovir
  Interventions: Behavioral: instructions and coaching
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: instructions and coaching — instructions and coaching or no intervention on the use and intake of ganciclovir
  Arms: 1

SUMMARY:
21 patients were randomised to receive instructions and coaching or no intervention on the use and intake of ganciclovir. Intake of medication was measured by an electronic pill box. The duration of the study was 100 days.

ELIGIBILITY:
Inclusion Criteria:

* men and women between 18 and 65 years old
* de novo kidney transplant patients
* patients who need CMV prophylaxis with ganciclovir during 3 months
* patients who gave informed consent after an oral explanation of the study

Exclusion Criteria:

* patients who are seronegative for CMV virus and who received a kidney from a CMV negative donor
* patients with a creatinin clearance of less than 10 ml/min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2001-05; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
relation between compliance of medication towards chemoprophylaxis and occurrence of CMV infection after kidney transplantation | weekly follow-up

SECONDARY OUTCOMES:
relation between compliance and the instructions which a patient gets about intake of medication | weekly follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Devolder, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- See also: Website University Hospital Ghent — http://www.uzgent.be